CLINICAL TRIAL: NCT01832675
Title: New Bupivacaine Lozenge as Topical Anesthesia Compared to Lidocaine Pharyngeal Spray Before Upper Gastrointestinal Endoscopy in Unsedated Patients
Brief Title: Clinical Trial With Bupivacaine Lozenges as Local Anaesthesia Under Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ove Andersen (Other)
Collaborators: Oracain II Aps (Unknown)
Responsible Party: Sponsor-Investigator, Ove Andersen, MD, PhD, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0056-22-21
Record Dates: First submitted 2013-01-04; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Application Site Discomfort
Keywords: Endoscopy; Anesthetics, Local; Bupivacaine; Lidocaine
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine lozenge (Active Comparator): The patients will either get lidocaine spray or bupivacaine lozenge as an anaesthetic drug before the upper gastroscopic endoscopy.
  Interventions: Drug: Bupivacaine lozenge
- Xylocain, cutaneous spray, solution (Active Comparator): The patients will either get lidocaine spray or bupivacaine lozenge as an anaesthetic drug before the upper gastroscopic endoscopy.
  Interventions: Drug: Xylocain, cutaneous spray, solution

INTERVENTIONS:
Drug: Xylocain, cutaneous spray, solution — 10 mg lidocaine/spray. The patient will be sprayed three times and get a maximal dose of 30 mg lidocaine just before the examination.
  Arms: Xylocain, cutaneous spray, solution
Drug: Bupivacaine lozenge — 25 mg bupivacaine/lozenge. The patient will get one lozenge 10-15 minutes before the examination.
  Arms: Bupivacaine lozenge

SUMMARY:
In this project the investigators want to compare a new anaesthetic method during upper gastroscopic endoscopy, compared to the traditional used method in a private clinic. The new method is a lozenge containing bupivacaine, and the traditional method is a lidocaine spray.

DETAILED DESCRIPTION:
The research group has previously conducted a clinical study with patients who underwent an UGE at the Department of Gastroenterology, Hvidovre University Hospital, Denmark, where the effect of a new lidocaine lozenge was compared to the lidocaine suspension that was used as standard treatment. The results showed that the lozenge increased the patient's acceptance of the gag reflexes, decreased the patient discomfort during UGE and thereby increased patient acceptance of the UGE. Furthermore, there was a significant improvement in assessment of taste and texture of the lozenge compared to the suspension. A study by Thanvi et al. has shown that it is difficult to obtain valid VAS scores when the patients are sedated, as it might cause amnesia and may impair the patient's ability to make an accurate assessment of the discomfort. Sedation were a limitation for the study conducted by the research group, because of impairment in the patients judgmental abilities. Furthermore a longer duration of the effect of the lozenge was requested. Therefore, the research group reformulated the lozenge and changed the active pharmaceutical ingredient (API) to bupivacaine. Bupivacaine is an amide as lidocaine, but has a longer anesthetic effect and is four times as potent as lidocaine. It would therefore be relevant to optimize the study design and perform a new clinical study with unsedated patients undergoing UGE, where the bupivacaine lozenge was tested.

The clinical study was performed in the private gastrointestinal (GI) clinic at Hvidovre, Denmark. Before the UGE was performed the patient was locally anesthetized in the pharynx with a lidocaine spray as a standard treatment.

The hypothesis was that a bupivacaine lozenge would reduce the patient experienced discomfort during UGE due to a better local anesthetic effect compared to lidocaine spray. Moreover it is hypothesized that the bupivacaine lozenge would be more patient friendly than the lidocaine spray because of a better taste masking according to lesser bitter taste and a pleasant mode of being anesthetized.

The aim of the study was to compare patient discomfort by two different local anesthetic methods. The standard treatment was a lidocaine pharyngeal spray and was compared to the experimental treatment a bupivacaine lozenge. The efficacy and acceptance of the treatments were also examined, as well as the taste of the anesthetics. Furthermore the patient's and endoscopist's assessment of the UGE was examined.

ELIGIBILITY:
Inclusion Criteria:

* Referral from personal doctor for the upper gastroscopic endoscopy
* Age between 18 and 80 year
* Able to speak, read and understand the danish language
* Must be informed orally and released a written consent and a signed authorization statement

Exclusion Criteria:

* Known allergy to bupivacaine or other local anesthetics of the amide type.
* Pregnancy - the patient will be asked if she uses sufficient contraception. When in doubt a pregnancy test will be performed.
* Breastfeeding
* Use of other medicine before the examination besides the experimental medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The patient experienced discomfort assessed on the Visual Analog Scale | Day 1
  The patient experienced discomfort during a upper gastroscopic endoscopy when using bupivacaine lozenge instead of lidocaine spray assessed on the Visual Analog Scale

SECONDARY OUTCOMES:
Patient evaluation of taste and texture on a 3 point scale. - The investigator's assessment of the study by answering the questionnaire. | Day 1
  Patient evaluation of taste and texture of the lozenge or the spray on a 3 point scale.
Endoscopist evaluation on a 4 point scale. | Day 1
  The endoscopist evaluate the difficulty of the upper gastrointestinal endoscopy on a 4 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kaare Nielsen, MD, Principal Investigator — Kirurgisk Klinik Hvidovre
Locations (1):
- Kirurgisk Klinik Hvidovre, Hvidovre, Denmark